CLINICAL TRIAL: NCT06229912
Title: A Phase II Study of the Menin Inhibitor Revumenib in Leukemia Associated With Upregulation of HOX Genes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0660; NCI-2024-00534 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Leukemia; HOX Gene
MeSH Terms: conditions — Leukemia | interventions — revumenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Participants found to be eligible to take part in this study, will take revumenib 2 times a day (each dose about 12 hours apart), every day of each 28-day study cycle.
  Interventions: Drug: Revumenib

INTERVENTIONS:
Drug: Revumenib — Given by PO
  Other Names: SNDX- 5613

SUMMARY:
To learn if revumenib (also known as SNDX-5613) can help to control leukemias associated with an increase in expression of HOX genes.

DETAILED DESCRIPTION:
Primary Objectives

• To assess the efficacy of revumenib in leukemias associated with upregulation of HOX genes.

Secondary Objectives

* To assess rates of measurable residual disease (MRD) clearance, as assessed by multiparameter flow cytometry in participants who respond to treatment.
* To assess rates of cytogenetic remissions in participants with baseline cytogenetic abnormalities at diagnosis.
* To assess event-free survival (EFS), duration of response (DOR), and overall survival (OS) in participants with leukemia associated with upregulation of HOX following treatment with revumenib.

Exploratory Objectives

* To evaluate molecular and cellular markers that may be predictive of antitumor activity and/or resistance
* To evaluate HOX/MEIS1 expression as a biomarker of response.
* To assess the rate of mutations in the MEN1 gene as a mechanism of resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 years with weight ≥ 40Kg.
2. ECOG performance status of ≤ 2.
3. Relapsed or refractory acute leukemia, of either myeloid, lymphoid or mixed lineages, with genetic alterations associated with upregulation of HOX, as specified below:

   Alteration/Mutation - Cytogenetics KMT2A-PTD = Normal karyotype; NPM1-MLF1 = t(3;5)(q25;q34); NUP98r = 11p15 rearrangements; SET-NUP214 = t(9;9)(q34;q34); RUNX1-EVI1 = t(3;21)(q26;q22); MYST3-CREBBP = t(8;16)(p11;p13); CDX2-ETV6 = t(12;13)(p13;q12); CALM-AF10 = t(10;11)(p13;q14-21); MN1-ETV6 = t(12;22)(p13;q12); UBTF-TD = Normal karyotype
4. WBC must be below 25,000/ uL at time of enrollment. Participants may receive cytoreduction prior to enrollment.
5. Baseline ejection fraction must be > 40%.
6. Adequate hepatic function (direct bilirubin < 1.5x upper limit of normal (ULN) unless increase is due leukemic involvement, and AST and/or ALT < 3x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT < 5x ULN will be considered eligible).
7. Adequate renal function with an estimated glomerular filtration rate ≥ 60 mL/min based on local institutional practice for age-appropriate determination.
8. Participants or parent/guardian is willing and able to provide informed consent.
9. In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 14 days for cytotoxic or non-cytotoxic (immunotherapy agent(s), or an interval of 5 half-lives of the prior therapy. Oral hydroxyurea and/or cytarabine (up to 2 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the principal investigator (PI). Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted.
10. Women of childbearing potential must agree to adequate methods of contraception during the study and at least 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study and at least 3 months after the last treatment.

Exclusion Criteria:

1. Participants with any concurrent uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the participant at unacceptable risk of study treatment.
2. The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions (1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia. (2) use of hydroxyurea for participants with rapidly proliferative disease or for control of counts during differentiation syndrome. (3) use of steroids for treatment of differentiation syndrome.
3. Participants with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
4. Participants with concurrent active malignancy under treatment.
5. Known active hepatitis B (HBV) or hepatitis C (HCV) or human immunodeficiency virus (HIV) infections.
6. Female subjects who are pregnant or breast-feeding.
7. Participant has an active uncontrolled infection.
8. Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack.
9. QTc >450 msec for males and QTc >470 msec for females using the Fridericia Formula using an average of the 3 Screening EKGs.
10. History of or any concurrent condition, therapy, or laboratory abnormality that in the Investigator's opinion might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate.
11. Clinically active central nervous system (CNS) leukemia.
12. Participants on immunosuppressive therapy post-HSCT at the time of screening (must be off all systemic immunosuppression therapy for at least 2 weeks and calcineurin inhibitors for at least 4 weeks). The use of topical steroids for cutaneous graft-versus-host disease (GVHD) or stable systemic steroid doses less than or equal to 20 mg of prednisone (or equivalent) daily are permitted.
13. Participants with Grade > 2 active acute GVHD, moderate or severe limited chronic GVHD, or extensive chronic GVHD of any severity.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ghayas Issa, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org